CLINICAL TRIAL: NCT01740739
Title: Evaluation Using ClearView in Determining Association to the Cardiac Risk Factors (Cardiac-CV)
Brief Title: Evaluation Using ClearView in Determining Association to the Cardiac Risk Factors
Acronym: Cardiac-CV
Status: Suspended | Type: Observational
Why Stopped: Evaluating cohort for value
Sponsor: Epic Research & Diagnostics, Inc. (Industry)
Collaborators: Mission Internal Medical Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: EPIC-006
Record Dates: First submitted 2012-11-16; First posted 2012-12-04 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease
Keywords: Health Risk Appraisal; HCardiac Risk Factors
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Risk: Patients, as part of their standard of care, who are recommended for and who complete a test resulting in a Coronary Calcium Score, lipid test, hs-CRP and MPO result.

SUMMARY:
The objective of this study is to explore the relationship between the ClearView scan results and a variety of cardiovascular risk indicators such as the Coronary Calcium Score, Framingham Risk Factors, Reynolds Risk Score, and biomarkers of inflammation. The ClearView device is a bio-electrographic tool that may assist medical professionals in rapid assessment of the systemic origin of the patient's presenting symptom(s). The ClearView is a potentially valuable resource that may benefit a physician's office by offering expedited differentiation capabilities. The subsequent results have the potential to include more data that would allow rapid patient diagnosis, triage, and treatment; optimized precious resource expenditure (nursing, physician, etc.); lower costs to facility, patient and insurance company; and decreased office wait time.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male or Female
* Age range: 18 to 85
* Patients who are recommended for and who have had a cardiac CT study that produces a Coronary Calcium Score within 30 days prior to the ClearView Scan or plan to have the CT within 14 days after the ClearView Scan.
* Patients who have had a blood test resulting in hs-CRP, fasting lipid panel and MPO results within 6 months prior to the ClearView Scan or plan to have the tests done within 14 days after the ClearView Scan.
* The patient or legal representative is able to understand and provide signed consent for the procedure.

Exclusion Criteria:

* Patients with pacemakers or another implanted electrical device, such as an automatic internal cardiac defibrillator.

  * Patients connected to an electrical device that cannot be removed or temporarily powered off (i.e. monitor) during subject testing with the ClearView Device
  * Vulnerable populations
  * Patients actively being treated for cancer or with a previous diagnosis of cancer that required chemotherapy, radiation therapy or hormonal therapy.
  * Patients missing all or any part of a fingertip (excluding fingernail).
  * Patients with involuntary hand tremors /shaking of the hands that may prevent clear imaging.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and Women, as part of their standard or care, who are recommended for and who complete a test resulting in a Coronary Calcium Score, hs-CRP, and MPO result.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Association of ClearView scan with cardiovascular risk indicators | Single Study Vist, no follow-up.
  Statistical agreement will be assessed between the ClearView Response result and the results of the Corinary Calcium Score, Inflammatory biomarkers, lipid panel results and cardiovascular risk indicators as reported by the medical exam, on a per-subject basis.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Miyamoto, MD, Principal Investigator — Mission Internal Medical Group
Locations (1):
- Mission Internal Medical Group, Mission Viejo, California, United States